CLINICAL TRIAL: NCT02547207
Title: MultiPoint Pacing Mapping Study
Status: Terminated | Type: Observational
Why Stopped: Slow recruitment
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CR-13-004-EU-HF
Record Dates: First submitted 2015-05-07; First posted 2015-09-11 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to characterize left ventricular acute hemodynamic and electrical responses during cardiac resynchronization therapy (CRT) with different Multipoint Pacing (MPP) settings, and assess the relationship between electrical activation patterns and hemodynamic measurements during these pacing settings.

ELIGIBILITY:
Inclusion Criteria:

* Be scheduled to undergo or have received within the past 30 days an implant of a SJM (St. Jude Medical) MPP CRT-D system with approved standard indication by ESC (European Society of Cardiology) / EHRA (European Heart Rhythm Association) Guidelines
* Have the ability to provide informed consent for study participation and be willing and able to comply with the Clinical Investigation Plan (CIP) described evaluations and follow-up schedule
* Be in sinus rhythm

Exclusion Criteria:

* Complete AV (atrioventricular) block
* Permanent atrial fibrillation
* Have a recent myocardial infarction within 40 days prior to enrollment
* Have undergone cardiac surgery or coronary revascularization procedure within 3 months prior to enrollment or be scheduled for such procedures in the following 7 months
* Have had a recent CVA (cerebrovascular accident) or TIA (transient ischemic attack) within 3 months prior to enrollment
* Have had intravenous inotropic support in the last 30 days
* Be less than 18 years of age
* Be pregnant or plan to become pregnant over the next 7 months
* Have significant peripheral vascular disease
* Have LV thrombus
* Significant aortic valve disease or replacement
* Mitral valvular disease
* Contraindicated for Gadolinium contrast agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients meeting specific eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Left ventricular (LV) dP/dt Max (maximum change in pressure over time) in mmHg/s during different pacing settings | up to 30 days post-implant

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Leclercq, MD, PhD, Principal Investigator — University Hospital Rennes, Rennes, France
Locations (4):
- CHU Pontchaillou, Rennes, France
- Germany (2):
  - Kerckhoff-Klinik GmbH, Bad Nauheim
  - Herzzentrum Dresden Universitätsklinik, Dresden
- St. Thomas Hospital, London, United Kingdom